CLINICAL TRIAL: NCT05748925
Title: Study of the Cardio Renal Effects of SGLT2 Inhibitors Among Diabetic and Non-diabetic Lupus Nephritis Patients
Brief Title: Cardio Renal Effects of SGLT2 Inhibitors Among Lupus Nephritis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Nourelsabah Mohamed, Nephrology specialist at mansoura urology and nephrology center, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MD.21.10.550
Record Dates: First submitted 2023-02-18; First posted 2023-03-01 (Actual); Results first posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: SLE; Lupus Nephritis; SGLT2 Inhibitors
MeSH Terms: conditions — Lupus Nephritis | interventions — dapagliflozin

STUDY DESIGN:
Intervention Model Description: randomized controlled trial, It will include 100 patients with lupus nephritis, Diagnosis of glomerulonephritis was performed by renal biopsy, and all of the renal biopsies were carried out at urology and nephrology center.
  Patients with an estimated glomerular filtration rate (eGFR) >30 ml/min/1.73m2 will be randomized into two groups Study group will receive SGLT2i inhibitor as add on drug or replace another drug according to patient clinical situation, Dapagliflozin 10 mg and 25 mg will be used once daily with or without food.
  Control group will be maintained on placebo.
Who Masked: Participant, Care Provider
Masking Description: double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Active Comparator): study group: will receive SGLT2i as add on drug or replace another drug according to the patient clinical situation, Dapagliflozin 10 mg will be used once daily with or without food for one ye
  Interventions: Drug: dapagliflozin
- control group (Active Comparator): Control group: will receive placebo as add on drug once daily with or without food for one year.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: dapagliflozin — The patients will be randomized into two groups Study group: will receive SGLT2i as add on drug or replace another drug according to the patient clinical situation, Dapagliflozin 10 mg will be used once daily with or without food.
  Arms: study group
Drug: placebo — Control group: will be maintained on their medication
  Arms: control group

SUMMARY:
This study aims to assess sodium glucose linked transoprter inhibitors(SGT2i) role in regression of ongoing kidney and cardiac diseases among lupus nephritis patient either diabetic or non-diabetic under different immunosuppressive therapy.

The main objective of this study is to:

To compare use of sodium glucose linked transoprter inhibitors (SGLT2i) versus standard care in regression of chronic kidney disease in patient with lupus nephritis (LN).

To study the safety and efficacy of this drug group with use of immunosuppression and possible interaction.

Patients with an estimated glomerular filtration rate (eGFR) >30 ml/min/1.73m2 will be randomized into two groups Study group will receive SGLT2i inhibitor as add on drug or replace another drug according to patient clinical situation, Dapagliflozin 10 mg and 25 mg will be used once daily with or without food.

Control group will be maintained on placebo.We will follow up all patients for 12 months and compare their results.

DETAILED DESCRIPTION:
Study sitting:

Nephrology and renal transplant unit at urology and nephrology center in Mansoura University.

It will include 100 patients with lupus nephritis, Diagnosis of glomerulonephritis was performed by renal biopsy, and all of the renal biopsies were carried out at urology and nephrology center.

Patients with an estimated glomerular filtration rate (eGFR) >30 ml/min/1.73m2 will be randomized into two groups Study group will receive SGLT2i inhibitor as add on drug or replace another drug according to patient clinical situation, dapagliflozin 10 mg and 25 mg will be used once daily with or without food.

Control group will be maintained on placebo. The primary endpoint will be sustained decline in eGFR ≥50%, ESKD, or kidney or cardiovascular death We will follow up all patients for 12 months and compare their results.

2. Inclusion criteria: Patients aged more than 16 year. Willing to sign informed consent. Diagnosis of Systemic Lupus Erythematosus (SLE) according to american college of rheumatology (ACR) classification criteria.

Renal biopsy showed lupus nephritis. Patient with eGFR > 30 ml/min/1.73m2 by cockcroft-gault equation. 3. Exclusion criteria: Patients with eGFR <30 ml/min per 1.73 m2. Current pregnancy or lactation. Medical history of chronic disease (CLD, cancer, severe respiratory distress, gastrointestinal tract lesions).

Patients refusing to participate in the study or lost follow up. Evidence of urinary obstruction of difficulty in voiding at screening. Patients who are receiving high dose diuretics or combined Angiotensin converting enzymes inhibitors(ACEI) and Angiotensin II receptor blockers (ARBS).

Patients who have frequent hypotensive episode or systolic blood pressure (SBP) <100 mmHg.

Operational design:

Study Protocol:

Patients included in the study will treated with dapaglifilozin initiated at a total daily dosage of 10 mg/kg per day.

Study design:

Type of the study: randomized controlled study.

The following data will be gathered and evaluated for all patients:

I-before intervention:

Serum creatinine, Creatinine clearance. 24 hour urine protein, urine protein/creatinine ratio. Urine analysis. HBA1c. Hemoglobin (HGB). Uric acid and lipid profile. Lupus serology.

II-after intervention: All patients will be evaluated monthly regarding:

Serum creatinine, creatinine clearance. 24 hour proteinuria, protein/creatinine ratio. Fasting, random and postprandial glucose levels. calcineurin inhibitors (CNI) trough level if used. Urine analysis. HGB level. Uric acid, lipid profile. Lupus serology.

Cardiovascular assessment:

Echocardiogram. Atherosclerosis and vascular calcification incidence (NCCT model). Regular measurement of blood pressure each visit

ll patients will be evaluated at 12 month regarding:

1. erythropoetin level
2. Hepcidin level.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged more than 16 year.
* Willing to sign informed consent.
* Diagnosis of SLE according to EULAR/ACR classification criteria.
* Renal biopsy showed lupus nephritis.
* Patient with eGFR > 30 ml/min/1.73m2 by cockcroft-gault equation.

Exclusion Criteria:

* Patients with eGFR <30 ml/min per 1.73 m2.
* Current pregnancy or lactation.
* Medical history of chronic disease (CLD, cancer, severe respiratory distress, gastrointestinal tract lesions).
* Patients refusing to participate in the study or lost follow up.
* Evidence of urinary obstruction of difficulty in voiding at screening.
* Patients who are receiving high dose diuretics or combined ACEI, Angiotensin II receptor blockers (ARBS).
* Patients who have frequent hypotensive episode or SBP <100 mmHg.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Urology and Nephrology Center, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: Yes
all individual participant data (IPD) that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: 1 year

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Study Group | Control Group
Started | 42 | 42
Completed | 38 | 41
Not Completed | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Study Group | Control Group | Total
Number analyzed (Participants) | 38 | 41 | 79
Age, Customized [Mean (Standard Deviation); unit: years] | 38 (9.8) | 36.6 (9.6) | 37.3 (9.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 34 | 68
  Male | 4 | 7 | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body weight (Kg) [Mean (Standard Deviation); unit: kilograms (kg)] | 90 (15) | 78.9 (14) | 84.3 (15.7)
Body mass index [Mean (Standard Deviation); unit: kilograms per square meter (kg/m²)] | 33 (5.7) | 30.6 (10.5) | 31.9 (8.5)
Hypertension [Count of Participants; unit: Participants] | 38 | 37 | 75
Diabetes [Count of Participants; unit: Participants] | 11 | 7 | 18

OUTCOME MEASURES:

1. Primary Outcome: Effect of Dapagliflozin Compared to Placebo on Renal Function After One Year
Description: Effect of dapagliflozin compared to placebo on eGFR,24- hour urinary protein
Time Frame: one year
Measure: Mean (Standard Deviation); unit: mL/min/1.73 m²
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 38 | 41
mL/min/1.73 m²
  eGFR Baseline | 128 (59.7) | 114 (51)
  eGFR 12 months | 115.7 (48) | 100.3 (44.5)

2. Primary Outcome: Cardiovascular Assessment in Two Groups
Description: Coronary artery calcification will be measured using non-contrast computed tomography (NCCT). The Agatston score, a standardized method for quantifying coronary calcification, will be used to assess and compare baseline and 1-year follow-up measurements between the dapagliflozin and placebo groups.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 38 | 41
Participants
  Coronary calcification baseline | 11 | 3
  Coronary calcification 12 months | 11 | 1

3. Primary Outcome: Effect of Dapagliflozin Compared to Placebo on Erythropoietin Level
Description: Erythropoietin level will be measured in two groups before and after intervention
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: international units per liter (IU/L)
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 38 | 41
international units per liter (IU/L)
  Erythropoietin level baseline | 11.3 (1.4) | 11.6 (2.1)
  Erythropoietin level 12 months | 12.4 (3.5) | 12.8 (3.5)

4. Primary Outcome: Effect of Dapagliflozin Compared to Placebo on Hepcidin Level
Description: hepcidin level will be measured in two groups before and after intervention
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 38 | 41
nanograms per milliliter (ng/mL)
  Hepcidin level Baseline | 182 (76) | 198 (74)
  Hepcidin level12 months | 116 (15) | 128 (63)

5. Primary Outcome: Effect of Dapagliflozin Compared to Placebo on Renal Function
Description: Effect of dapagliflozin compared to placebo on 24- hour urinary protein after 1 year
Time Frame: 1 year
Measure: Median (Inter-Quartile Range); unit: grams per 24 hours (g/24 hours)
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 38 | 41
grams per 24 hours (g/24 hours)
  24- hour urinary protein baseline | 0.6 [0.07 to 3] | 0.5 [0.02 to 4]
  24- hour urinary protein 12months | 0.4 [0.06 to 3.6] | 0.5 [0.02 to 8]

6. Primary Outcome: Effect of Dapagliflozin Compared to Placebo on Renal Function
Description: Effect of Dapagliflozin Compared to Placebo on Renal Function on uric acid after 1 year
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 38 | 41
milligrams per deciliter (mg/dL)
  Uric acid baseline | 6.5 (1.7) | 6.2 (2.1)
  Uric acid 12 months | 5.8 (1.5) | 6.2 (1.8)

7. Secondary Outcome: Effect of Dapagliflozin Compared to Placebo on ECCHO Parameters
Description: ECCHO will be done before and after intervention
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: Percentage (%)
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 38 | 41
Percentage (%)
  EF baseline | 64.6 (5.4) | 64.4 (9.3)
  EF 12months | 64.9 (5.2) | 65.8 (5.8)

8. Secondary Outcome: Effect of Dapagliflozin Compared to Placebo on Body Weight
Description: body weight will be assessed throughout the study
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: kilo gram
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 38 | 41
kilo gram
  body weight baseline | 90 (15.4) | 78.9 (14.1)
  body weight 12months | 87 (14) | 77.9 (14.3)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Study Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/41
Serious Adverse Events (participants affected / at risk) | 7/38 | 3/41
Other Adverse Events (participants affected / at risk) | 4/38 | 2/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Group (N=38) | Control Group (N=41)
AKI (Renal and urinary disorders) | 7 (7) | 3 (3) — AKI after intervention
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Group (N=38) | Control Group (N=41)
UTI (Infections and infestations) | 4 (4) | 2 (2) — UTI after intervention

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2024-05-11): https://cdn.clinicaltrials.gov/large-docs/25/NCT05748925/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-11): https://cdn.clinicaltrials.gov/large-docs/25/NCT05748925/SAP_001.pdf